CLINICAL TRIAL: NCT01957072
Title: Pilot Study of Behavioural Intervention for Nutrition in Cystic Fibrosis
Acronym: PIN-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STH17327; IRAS Project ID 139047 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Nutrition; Weight; BMI; Behaviour change
MeSH Terms: conditions — Cystic Fibrosis; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behaviour change intervention (Experimental): Intensive behaviour change intervention for 3 months, followed by a maintenance phase for 3 months
  Interventions: Behavioral: Behaviour change intervention
- Wait-list Control (Other): Usual care for 3 months, followed by intensive behaviour change intervention for 3 months
  Interventions: Behavioral: Behaviour change intervention

INTERVENTIONS:
Behavioral: Behaviour change intervention — The behaviour change intervention consists of
  1. feedback via a web-based food diary
  2. 'coaching' with problem-solving and implementation plans
  The intensive intervention phase consists of 2 home visits, 8 telephone calls and 6 reminder emails.
  The maintenance phase consists of 3 telephone calls and 4 reminder emails.

SUMMARY:
Cystic Fibrosis (CF) is a lifelong condition which causes the lungs and digestive system to become clogged with thick, sticky mucus. This leads to recurrent lung infections and reduced nutrients absorption from food. The average age at death is 26 years, usually from respiratory failure. Nonetheless, the nutritional status of people with CF (PWCF) is important help them live healthier and longer.

It is recommended that adult with CF achieve a BMI of 23 for males and 22 for females. However, fewer than 50% adult with CF achieved that target BMI despite effective nutritional support to help support weight gain. There is a clear need for a behavioural intervention that can help PWCF use the available nutritional support.

This is a feasibility study to try out a multi-component behavioural intervention. The intervention is designed to help PWCF use their nutritional support to gain weight. It will focus on testing the methods and procedures to be used on a larger scale, improving the behavioural intervention and estimating the how many people are needed for the larger trial.

All eligible 75 PWCF in Sheffield will be invited to participate. The investigators anticipate recruiting 30 participants. Participants will be divided into two groups. The first group receive the behavioural intervention immediately. The second group receive the intervention after 3 months. All participants will be followed up for 6 months. Data will be collected every 6 weeks during clinic reviews.

These two groups will be compared against each other to estimate the potential impact of the behavioural intervention. The investigators will also interview some of the participants at the end of the study period to improve the intervention and the study processes based on participant feedback.

The investigators hypothesised that this study will recruit around 30 participants, around 80% of the participants will complete the study, a single full-time investigator can deliver the intervention to 15 participants over 3 months and data collection will be thorough (with less than 5% missing data). The investigators also hypothesised that this feasibility study will help improve the intervention and help the design of a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* adult people with CF looked after at the Sheffield Adult CF Unit
* best BMI of < 23 for males and < 22 for females between Oct '12 and Oct '13

Exclusion Criteria:

* patients in the palliative phase of disease
* patients who are pregnant
* patients who have no capacity to consent to participate in the study
* patients who have no IT facilities to use the web-based food diary
* patients who are unable to communicate by telephone for coaching

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who accepted invitation to participate as a marker of feasibility | 4 weeks
Proportion of people with CF who are randomised into the study after accepting the invitation to participate, as a marker of feasibility | 4 weeks

SECONDARY OUTCOMES:
Participants' opinion about the behavioural intervention | 6 months
Participant attrition rate and phases of study whereby the attrition occurs | 6 months
Participants' opinion about the study processes | 6 months
Participants' suggestions for further improvement of the intervention and study processes | 6 months
Proportion of adults who fulfils the BMI criteria for recruitment with IT facilities | 2 weeks
Resources needed by the investigators to deliver the intervention | 6 months
Proportion of days with missing nutritional data, as a marker for feasibility | 6 months
  Participants are requested to fill in their nutritional intake daily on a web-based food diary. The investigators are interested to find out what the proportion of such data will be missing to determine the feasibility of collecting data with the web-based food diary.

OTHER OUTCOMES:
Body mass index | 6 months
  Unit is kg/m2
Weight | 6 months
  unit is kg
Beliefs about Medicines Questionnaire (BMQ) score | 6 months
  As a marker of patients' perception of their treatment
The mean Self-Report Behavioural Automaticity Index (SRBAI) score | 6 months
  As a marker of habit formation

CONTACTS AND LOCATIONS:
Overall Officials: Martin J Wildman, PhD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Northern General Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom